CLINICAL TRIAL: NCT04809779
Title: PD-1 Inhibitor Sintilimab Concurrent With Epirubicin Cyclophosphamide and Nab-paclitaxel as Neoadjuvant Therapy for Triple Negative Breast Cancer
Brief Title: PD-1 Inhibitor Concurrent With Chemotherapy as Neoadjuvant Therapy for TNBC
Acronym: NeoPD1TNBC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ying Lin, Vice Director, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020466
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sintilimab (Experimental)
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — The PD-1 inhibitor Sintilimab 200mg for intravenous (IV) administration will be given together with three-week epirubincin, cyclophosphamide (EC) × 4 treatments from the second cycle followed by weekly nab-paclitaxel x12 treatments or three-week nab-paclitaxel x4 treatments.

SUMMARY:
The purpose of the study is to address the following hypotheses: the PD-1 inhibitor Sintilimab 200mg for intravenous (IV) administration will be given together with three-week epirubincin, cyclophosphamide (EC) × 4 treatments from the second cycle followed by weekly nab-paclitaxel x12 treatments or three-week nab-paclitaxel x4 treatments. This regimen will induce higher pathologic complete response (pCR) rate in triple negative breast cancer than historical pCR rates (30-40%) observed with chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histologically confirmed stage I-III, ER, PR and HER2 negative invasive breast cancer as defined by the ASCO CAP guidelines for whom systemic chemotherapy would be indicated based on physician judgment following standard NCCN practice guidelines.

Exclusion Criteria:

* Patients for whom anthracycline, nab-paclitaxel or antibody therapies are contraindicated.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) | 21 weeks
  Pathologic response will be assessed in the surgically resected cancer and lymph nodes after completion of all chemotherapy by the local pathologist as part of routine care. Pathologic complete response is defined as no invasive cancer in the resected breast tissue and lymph nodes (ypT0/Tis, ypN0).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, China